CLINICAL TRIAL: NCT04823013
Title: Comparison of High Power Pain Threshold Ultrasound and Ischemic Compression Techniques for the Treatment of Latent Myofascial Trigger Points: A Randomized Controlled Study
Brief Title: Comparison of High Power Pain Threshold Ultrasound and Ischemic Compression Techniques for Treatment of Trigger Points
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Gamze Pala, Research Assistant, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B.30.2.AYD
Record Dates: First submitted 2021-03-24; First posted 2021-03-30 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Trigger Point Pain, Myofascial
Keywords: high power pain threshold ultrasound; ischemic compression; pain; trigger points; pain pressure threshold
MeSH Terms: conditions — Myofascial Pain Syndromes; Pain | interventions — Acupressure

STUDY DESIGN:
Intervention Model Description: Participants in HPPT-US 1 group received the HPPT-US treatment (n=52). The intensity was gradually increased from 0.5 W/cm² to the pain threshold level at which the patient verbally reported the pain. The therapist kept the intensity at that level for 5 s, and then moved the US transducer in a circle without the change of the intensity for 15 s. The procedure was repeated 3 times. Participants in HPPT-US 2 group also received the HPPT-US treatment (n=57). The intensity was gradually increased from 0.5 W/cm² to the pain threshold level at which the patient verbally reported the pain. The therapist kept the intensity at that level for 5 s, then reduced the dose half and moved the US transducer in a circle for 15 s. The procedure was repeated 3 times.Participants in IC group received ischemic compression therapy (n=44). The duration for each trigger points was 1 minute.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- high power pain threshold ultrasound which the dose was kept constant group (HPPT-US 1) (Experimental): Participants in HPPT-US 1 group received one session of HPPT-US treatment which the dose was kept constant. The technique delivers sound waves directly to the myofascial trigger points and results in immediate pain relief.
  Interventions: Other: high power pain threshold ultrasound which the dose was kept constant
- high power pain threshold ultrasound which the dose reduced to one half group (HPPT-US 2) (Experimental): Participants in HPPT-US 2 group received one session of HPPT-US treatment which the dose reduced to one half. The technique delivers sound waves directly to the myofascial trigger points and results in immediate pain relief.
  Interventions: Other: high power pain threshold ultrasound which the dose reduced to one half
- ischemic compression group (Experimental): Participants in IC group received one session of ischemic compression therapy. Ischemic compression is a therapy technique used in manual therapy, where blockage of blood in an area of the body is deliberately made, so that a resurgence of local blood flow will occur upon release.
  Interventions: Other: ischemic compression

INTERVENTIONS:
Other: high power pain threshold ultrasound which the dose was kept constant — Participants in HPPT-US 1 group received the HPPT-US treatment. The intensity was gradually increased from 0.5 W/cm² to the pain threshold level at which the patient verbally reported the pain. The therapist kept the intensity at that level for 5 s, and then moved the US transducer in a circle without the change of the intensity for 15 s. The procedure was repeated 3 times. The patients were asked whether serious pain or any abnormal sensation was felt during HPPT-US. The intensity was varied from 0.5 to 1.2 W/ cm².
  Arms: high power pain threshold ultrasound which the dose was kept constant group (HPPT-US 1)
Other: high power pain threshold ultrasound which the dose reduced to one half — Participants in HPPT-US 2 group also received the HPPT-US treatment. The intensity was gradually increased from 0.5 W/cm² to the pain threshold level at which the patient verbally reported the pain. The therapist kept the intensity at that level for 5 s, then reduced the dose half and moved the US transducer in a circle for 15 s. The procedure was repeated 3 times. The patients were asked whether serious pain or any abnormal sensation was felt during HPPT-US. The intensity was varied from 0.5 to 1.2 W/ cm².
  Arms: high power pain threshold ultrasound which the dose reduced to one half group (HPPT-US 2)
Other: ischemic compression — Participants in IC group received ischemic compression therapy. The technique was applied in the sitting position to participants. Ischemic compression was performed by compressing trigger points identified by palpation with tolerable intensity using thumb. The duration for each trigger points was 1 minute. Then the muscle containing the trigger point was applied intramuscular stretching for 30 seconds by therapist
  Arms: ischemic compression group

SUMMARY:
This study aimed to compare the efficacy of ischemic compression and two different application methods of high power pain threshold ultrasound techniques on latent trigger point treatment. Asymptomatic subjects divided into three groups. First group took high power pain threshold ultrasound in which the intensity is kept constant at the pain level; second group took high power pain threshold ultrasound which the intensity is kept constant at half the pain level and third group took ischemic compression. All participants were asked to complete the questionnaires, which assessed pain, psychological factors and disability before treatment, after 1 week and 1 month follow-up. After each participants completed the questionnaire, the physical therapist evaluated the MTrPs. MTrPs assessment was performed before treatment, immediately after treatment, after 1 week and 1 month follow-up.

DETAILED DESCRIPTION:
Myofascial trigger points have been defined as discrete and hyperirritable areas located within a taut band of skeletal muscle or fascia which when compressed produce pain, tenderness, dysfunction and autonomic phenomena. The treatment techniques aimed to return the fiber groups affected by myofascial trigger points to their normal length and endplates to their normal function. Although both ischemic compression and two different application methods of high power pain threshold ultrasound techniques are effective methods in the treatment of trigger points , there are no studies showing which technique is more effective. It is aimed to to compare the efficacy of ischemic compression and two different application methods of high power pain threshold ultrasound techniques on myofascial trigger point treatment.

ELIGIBILITY:
Inclusion Criteria:

1. being aged between 18-50
2. the presence of a minimum of 3 latent trigger points in Upper Trapezius, Levator Scapulae, Supraspinatus, Infraspinatus, Deltoid Anterior, Pectoralis Major, Pectoralis Minor muscles
3. no health problems
4. signed the voluntary consent form

Exclusion Criteria:

1. have a neck, spine or shoulder injury in the last 6 months
2. continued neck and back pain in the last 6 months
3. having a skin disease that may affect upper extremity assessment
4. malign and benign tumors
5. pain relief medication
6. having psychiatric treatment. -

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 153 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
Pain intensity | Pain intensity was measured using visual analog scale (VAS) before the treatment (0-10 numeric pain rating scale, with 0 indicating no pain and 10 severe pain)
  Pain intensity is of valuable diagnostic information, and we ask patients to evaluate how strong their pain feels
Beck Depression Inventory | Depression was assessed using the Beck Depression Inventory (BDI) before the treatment. BDI comprises 21 items, each of which is rated between 0 and 3 on a 4-point Likert Scale. The total score ranges from 0 to 63 points.
  Depression is a constant feeling of sadness and loss of interest, which stops you doing your normal activities.
Neck Pain and Disability Scale | Disability was evaluated by Neck Pain and Disability Scale (NPAD) before the treatment. The scale progresses from 0 to 5, increasing the limitation. the total NPAD score, which ranges from 0 to 100 points.
  A disability is any condition of the body or mind that makes it more difficult for the person with the condition to do certain activities (activity limitation) and interact with the world around them.
Myofascial trigger points assessment | The MTrPs assesment was made with palpation by the physical therapist. The therapist used an algometer. The number of MTrPs and pain pressure threshold values were evaluated before treatment. PPT is a safe outcome measure to evaluate pain sensitivity.
  Myofascial trigger points (MTrPs) have been defined as discrete and hyperirritable areas located within a taut band of skeletal muscle or fascia which when compressed produce pain, tenderness, dysfunction and autonomic phenomena
Myofascial trigger points assessment | The MTrPs assesment was made with palpation by the physical therapist. The therapist used an algometer. The number of MTrPs and pain pressure threshold values were evaluated immediately after the treatment.
  Myofascial trigger points (MTrPs) have been defined as discrete and hyperirritable areas located within a taut band of skeletal muscle or fascia which when compressed produce pain, tenderness, dysfunction and autonomic phenomena
Pain intensity | Pain intensity was measured using visual analog scale (VAS) at one week after the treatment (0-10 numeric pain rating scale, with 0 indicating no pain and 10 severe pain)
  Pain intensity is of valuable diagnostic information, and we ask patients to evaluate how strong their pain feels
Beck Depression Inventory | Depression was assessed using the Beck Depression Inventory (BDI) at one week after the treatment. BDI comprises 21 items, each of which is rated between 0 and 3 on a 4-point Likert Scale. The total score ranges from 0 to 63 points.
  Depression is a constant feeling of sadness and loss of interest, which stops you doing your normal activities.
Neck Pain and Disability Scale | Disability was evaluated by Neck Pain and Disability Scale (NPAD) at one week after the treatment. The scale progresses from 0 to 5, increasing the limitation. the total NPAD score, which ranges from 0 to 100 points.
  A disability is any condition of the body or mind that makes it more difficult for the person with the condition to do certain activities (activity limitation) and interact with the world around them.
Myofascial trigger points assessment | The MTrPs assesment was made with palpation by the physical therapist. The therapist used an algometer. Pain pressure threshold values were evaluated at one week after the treatment.
  Myofascial trigger points (MTrPs) have been defined as discrete and hyperirritable areas located within a taut band of skeletal muscle or fascia which when compressed produce pain, tenderness, dysfunction and autonomic phenomena
Pain intensity | Pain intensity was measured using visual analog scale (VAS) at one month after the treatment (0-10 numeric pain rating scale, with 0 indicating no pain and 10 severe pain)
  Pain intensity is of valuable diagnostic information, and we ask patients to evaluate how strong their pain feels
Beck Depression Inventory | Depression was assessed using the Beck Depression Inventory (BDI) at one month after the treatment. BDI comprises 21 items, each of which is rated between 0 and 3 on a 4-point Likert Scale. The total score ranges from 0 to 63 points.
  Depression is a constant feeling of sadness and loss of interest, which stops you doing your normal activities.
Neck Pain and Disability Scale | Disability was evaluated by Neck Pain and Disability Scale (NPAD) at one month after the treatment. The scale progresses from 0 to 5, increasing the limitation. the total NPAD score, which ranges from 0 to 100 points.
  A disability is any condition of the body or mind that makes it more difficult for the person with the condition to do certain activities (activity limitation) and interact with the world around them.
Myofascial trigger points assessment | The MTrPs assesment was made with palpation by the physical therapist. The therapist used an algometer. Pain pressure threshold values were evaluated at one month after the treatment.
  Myofascial trigger points (MTrPs) have been defined as discrete and hyperirritable areas located within a taut band of skeletal muscle or fascia which when compressed produce pain, tenderness, dysfunction and autonomic phenomena

CONTACTS AND LOCATIONS:
Overall Officials: Gamze G Pala, PhD, Principal Investigator — Istanbul Aydın University; Ebru Kaya Mutlu, Assoc.Prof., Principal Investigator — Istanbul University - Cerrahpasa; Hanifegül Taşkıran, Prof., Principal Investigator — Istanbul Aydın University
Locations (1):
- Istanbul Aydın University, Istanbul, Halit Aydın Kampüsü No:38 Küçükçekmece, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alvarez DJ, Rockwell PG. Trigger points: diagnosis and management. Am Fam Physician. 2002 Feb 15;65(4):653-60. PMID 11871683
- [Background] Vernon H, Schneider M. Chiropractic management of myofascial trigger points and myofascial pain syndrome: a systematic review of the literature. J Manipulative Physiol Ther. 2009 Jan;32(1):14-24. doi: 10.1016/j.jmpt.2008.06.012. PMID 19121461
- [Background] Unalan H, Majlesi J, Aydin FY, Palamar D. Comparison of high-power pain threshold ultrasound therapy with local injection in the treatment of active myofascial trigger points of the upper trapezius muscle. Arch Phys Med Rehabil. 2011 Apr;92(4):657-62. doi: 10.1016/j.apmr.2010.11.030. PMID 21440713